CLINICAL TRIAL: NCT04700722
Title: Cutaneous Phosphorlyated α-synuclein Detection as a Biomarker of Synucleinopathy
Brief Title: Synuclein-One Study
Status: Completed | Type: Observational
Sponsor: CND Life Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CND-100
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease; Multiple System Atrophy; Dementia With Lewy Bodies; Pure Autonomic Failure
Keywords: Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Lewy Body Disease; Pure Autonomic Failure; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Skin Biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Parkinson's disease: Looking for 105 patients with a clinically established diagnosis of Parkinson's disease between 40-99 years of age.
  Interventions: Diagnostic Test: Skin Biopsy
- Multiple System Atrophy: Looking for 40 patients with a clinically established diagnosis of Multiple System Atrophy between 40-99 years of age.
  Interventions: Diagnostic Test: Skin Biopsy
- Dementia with Lewy bodies: Looking for 95 patients with a clinically established diagnosis of Dementia with Lewy bodies between 40-99 years of age.
  Interventions: Diagnostic Test: Skin Biopsy
- Pure Autonomic Failure: Looking for 60 patients with a clinically established diagnosis of Pure Autonomic Failure between 40-99 years of age.
  Interventions: Diagnostic Test: Skin Biopsy
- Healthy Controls: No history of clinical or symptoms suggestive of Parkinson's disease, Multiple System Atrophy, Dementia with Lewy bodies or Pure Autonomic Failure between 40-99 years of age.
  Interventions: Diagnostic Test: Skin Biopsy

INTERVENTIONS:
Diagnostic Test: Skin Biopsy — Test accuracy and precision of skin biopsy detection of phosphorylated α-synuclein, define sensitivity and specificity of skin biopsy detection of phosphorylated α-synuclein deposition for the diagnosis of synucleinopathies and to differentiate between the synucleinopathies by quantitative measurement of phosphorylated α-synuclein with skin biopsies.

SUMMARY:
The Synuclein-One Study will be evaluating α-synuclein in patients with Parkinson's disease, Multiple System Atrophy, Dementia with Lewy bodies and Pure Autonomic Failure. Using a simple diagnostic test will improve clinical accuracy in diagnosing, earlier diagnosis, and distinguish between neurodegenerative diseases.

DETAILED DESCRIPTION:
Phosphorylated α-synuclein pathology in the diagnosis of synucleinopathies through qualitative and quantitative measurements of cutaneous phosphorylated α-synuclein in patients with Parkinson's disease, Multiple System Atrophy, Dementia with Lewy bodies and Pure Autonomic Failure. An effective tissue biomarker will provide an accurate diagnosis of α-synuclein in clinical practice, will differentiate between synucleinopathies, enable assessment of target engagement in the development of disease modifying and neuroprotective therapies and accelerate the development of neuroprotective and disease modifying therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 40-99 years of age
* Prior clinical diagnosis of Parkinson's disease, Multiple System Atrophy, Dementia with Lewy bodies or Pure Autonomic Failure
* Health Subjects, no history of clinical or symptoms suggestive with synucleinopathy

Exclusion Criteria:

* Clinical evidence of severe vascular disease (history of ulceration, poor wound healing, vascular claudication)
* Clinically active coronary artery or cerebrovascular disease
* Current smoker or alcoholism
* History of allergic reaction to local anesthesia for skin biopsies
* Use of blood thinners (aspirin or Plavix alone is allowed)
* Significantly impaired wound healing or history of scarring or keloid formation
* Healthy individuals or individuals with synucleinopathy is disease may be explained by other causes: recent history of encephalitis, Cortical dementia of Alzheimer's type, Whipple's disease, toxin exposure, repeated head injury and stepwise disease progression suggestive of vascular etiology

Ages: 40 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible men and women, age 40-99 years, will undergo a screening evaluation that includes a thorough medical history, physical and neurologic exam, orthostatic vitals, questionnaires and skin biopsy completed in one visit.
Sampling Method: Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Primary Outcome 1 | 2 years
  To define test accuracy and precision of skin biopsy detection of phosphorylated α-synuclein.
Primary Outcome 2 | 2 years
  To define sensitivity and specificity of skin biopsy detection of phosphorylated α-synuclein.
Primary Outcome 3 | 2 years
  To differentiate between the synucleinopathies by quantitative measurement of phosphorylated α-synuclein with skin biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Levine, MD, Principal Investigator — CND Life Sciences: www.cndlifesciences.com
Locations (23):
- United States (23):
  - MD First Research, Chandler, Arizona
  - CND Life Sciences, Phoenix, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - The Neuro Center, Carlsbad, California
  - Providence St. John's Health, Santa Monica, California
  - Rocky Mountain Movement Disorders Center, PC, Englewood, Colorado
  - Aventura Neurology, Aventura, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - UF College of Medicine, Gainesville, Florida
  - Parkinson's Disease Treatment Center SWFL, Port Charlotte, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Lahey Health, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NYU Medical Center, New York, New York
  - SouthShore Neurologic, Patchogue, New York
  - Duke University Medical Center, Durham, North Carolina
  - Providence Brain & Spine Institute, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UTSouthwestern, Dallas, Texas
  - Texas Movement Disorders Specialists, Georgetown, Texas
  - Evergreen Health, Kirkland, Washington
  - Swedish Neuroscience Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with researchers that are involved in the study.

REFERENCES:
- [Derived] Gibbons CH, Levine T, Adler CH, Bellaire B, Wang N, Agarwal P, Aldridge GM, Barboi A, Claassen D, Evidente VGH, Galasko D, Gonzalez-Duarte A, Gil R, Gudesblatt M, Isaacson SH, Kaufmann H, Khemani P, Kumar R, Lamotte G, Liu AJ, McFarland NR, Miglis MG, Reynolds A, Sahagian GA, Saint-Hilaire MH, Schwartzbard JB, Singer W, Soileau MJ, Vernino S, Millar Vernetti P, Yerstein O, Freeman R. Cutaneous Phosphorylated Alpha-Synuclein in Lewy Body Dementia. Ann Clin Transl Neurol. 2025 Dec 25. doi: 10.1002/acn3.70291. Online ahead of print. PMID 41449577
- [Derived] Gibbons CH, Freeman R, Bellaire B, Adler CH, Moore D, Levine T. Synuclein-One study: skin biopsy detection of phosphorylated alpha-synuclein for diagnosis of synucleinopathies. Biomark Med. 2022 May;16(7):499-509. doi: 10.2217/bmm-2021-0646. Epub 2022 Mar 11. PMID 35272481